CLINICAL TRIAL: NCT06245096
Title: Researching and Improving Psychotherapy Techniques in Interventions for DEpression (RIPTIDE)
Brief Title: Evaluating Process of Change in Cognitive Behavioral Therapy and Acceptance and Commitment Therapy for Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Iony Ezawa, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-23-01077
Record Dates: First submitted 2024-01-24; First posted 2024-02-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Over 8 sessions, clients learn techniques to challenge and change maladaptive thought and behavioral patterns
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Acceptance and Commitment Therapy (Active Comparator): Over 8 sessions, clients learn techniques to accept their negative internal experiences and commit to action in line with their values
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Sessions will focus on skills such as behavioral activation, mood tracking, identifying and reframing automatic thoughts, assertion training and smart goals.
  Arms: Cognitive Behavioral Therapy
Behavioral: Acceptance and Commitment Therapy — Sessions will focus on skills such as mindfulness, acceptance and willingness training, values clarification, committed action, defusion, and self-as-context.
  Arms: Acceptance and Commitment Therapy

SUMMARY:
This study will compare two psychological treatments for major depressive disorder (MDD): cognitive-behavioral therapy (CBT) and acceptance and commitment therapy (ACT). Both treatments are well-studied and supported by evidence as effective options for people experiencing depression. These treatments will be delivered in an online group format via Zoom.

The study will enroll up to 100 participants with depression. Half of the participants will receive online group CBT and half will receive online group ACT. There will be up to 10 members in each group. For both conditions, treatment will be provided over 8 weeks, with a 6-month follow-up period. Enrollment will be ongoing and groups will occur simultaneously.

Potential participants are asked to complete an initial screening and an intake evaluation to determine eligibility. They will then receive 8-weeks of treatment. Participants will complete self-report questionnaires throughout their time in the study.

DETAILED DESCRIPTION:
Some of the most powerful tools to combat depression come in the form of psychotherapies, including Cognitive Behavioral Therapy (CBT) and Acceptance and Commitment Therapy (ACT). While both treatments have been found to be generally effective in treating depression, they take fundamentally different treatment approaches. In CBT, clients learn techniques to challenge and change maladaptive thought and behavioral patterns. In ACT, clients learn techniques to accept their negative internal experiences and commit to action in line with their values. Despite being among the most effective treatments for depression, both CBT and ACT have a response rate of about only 50%. It is believe there are two key reasons investigators have not been able to improve these response rates. First, very little is known about which specific therapeutic skills are effective in these treatment packages. For example, do cognitive or behavioral change skills lead to therapeutic change in CBT? In ACT, do acceptance or change skills lead to therapeutic change? Second, it is not known which specific treatments or therapeutic skills work better for different individuals. Every individual has diverse needs, and therefore individuals may benefit differently from different treatment packages or from specific skills within each package.

Therefore, investigators plan to run a randomized controlled trial comparing CBT and ACT for depression in order to investigate which specific therapeutic skills are effective in these treatment packages. This approach will also allow investigators to identify predictors of differential response to treatment packages and specific treatment skills.

Upon joining the study, participants are asked to complete surveys for one week prior to starting treatment and again for one week once treatment is completed. During treatment, they are asked to complete surveys throughout the 8 weeks of therapy. Following the 8-week treatment, participants are asked to complete monthly follow-up surveys for 6 months.

There are three main objectives in this study. The first is to compare processes of change across the two treatments (i.e., what works in specific treatments?). The second is to determine client variables that predict differential treatment response (i.e., which treatment works best for a given client?). The third is to evaluate potential moderators of differential response to any specific skills across the treatments (i.e., which specific therapy skill works best for a given client?)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depressive disorder (MDD) according to DSM-V criteria (APA, 2013)
* 18 years of age or older
* access to a private location with a stable internet connection and a working video camera
* lives in California
* able to understand and speak English
* able and willing to give informed consent

Exclusion Criteria:

* current diagnosis other than MDD if it constitutes the predominant aspect of the clinical presentation and if it requires treatment other than that being offered
* clear indication of secondary gain (e.g., court ordered treatment)
* current suicide risk or significant intentional self-harm in the last six months sufficient to preclude treatment on an outpatient basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Chain of Change Treatment Diary (ChaCha-TD) | Three days per week during the eight-week course of treatment at 8 p.m. on preselected days.
  The ChaCha-TD designed by our research group assesses participants' affect, symptoms, quality of life, significant life events, skills use, and mechanisms of treatment change in daily life.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Questionnaire (GAD-7) | Intake, Post-treatment (8 weeks)
  The GAD-7 (Spitzer et al., 2006) is a seven-item self-report measure of anxiety symptom severity.
WHO Quality of Life-Brief (WHOQOL-BREF) | Intake, Post-treatment (8-weeks), and follow-up (6-months)
  The WHOQOL-BREF (WHOQOL Group; 1998) is a 26-item self-report measure that evaluates four dimensions of quality of life (physical health, psychological health, social relationships, environment. Each item ranges from 1-5 and items are summed upon completing the measure. Higher scores indicate greater satisfaction with quality of life.
Positive and Negative Affect Schedule (PANAS) | Intake, Post-treatment (8-weeks), and follow-up (6-months)
  The PANAS (Watson et al., 1988) is a 20-item scale that assesses the extent to which participants are experiencing different positive and negative emotions in the present moment. 10-items assess positive emotions and 10-items assess negative emotions. Items range from 1-5 and are summed based on the valence of the emotion. Higher scores indicate more salient experiences of affect.
Patient Health Questionnaire (PHQ-9) | Intake, Post-treatment (8-weeks), and follow-up (6-months)
  The PHQ-9 (Kroenke et al., 2001) is a 9-item self-report scale that measures depressive symptom severity. Each item ranges from 0-3 and items are summed upon completing the measures. Higher scores indicate greater depression symptom severity.
Discrimination-Related Vigilance Scale (DRVS) | Intake, Post-treatment (8-weeks)
  The DRVS (Williams, unpublished; and first published by Clark et al., 2006) is a 6-item measure of heightened vigilance in response to experiences of racial discrimination. This scale will be asked as a follow-up to the Brief PEDQ- CV to assess the extent to which the client is vigilant in their surroundings because of previous discrimination they experienced.
Valuing Questionnaire (VQ) | Intake, Post-treatment (8 weeks)
  The VQ (Smout et al., 2014) is a 10-item self-report measure that assesses the extent of personal values enactment during the past week.
Automatic Thoughts Questionnaire (ATQ) | Intake, Post-treatment (8 weeks)
  The ATQ (adapted from Hollon & Kendall, 1980) is a 30- item self-report checklist measure of common automatic thoughts participants may or may not have experienced in the past two weeks.
Emotion Regulation Questionnaire (ERQ) | Intake, Post-treatment (8 weeks)
  The ERQ (Gross & John, 2003) is a 10-item self-report measure of two emotion regulation strategies, cognitive reappraisal and expressive suppression.
Positive Valence Systems Scale (PVSS-21) | Intake, Post-treatment (8 weeks)
  The PVSS-21 (Khazanov et al,. 2020 ) is a self-report scale assessing the National Institute of Mental Health Research Domain Criteria Positive Valence Systems constructs (e.g., reward anticipation and initial reward responsiveness).
Multidimensional Scale of Perceived Social Support (MSPSS) | Intake, Post-treatment (8 weeks)
  The MSPSS (Zimet et al., 1988) is a 12-item measure of perceived adequacy of social support from family, friends, and significant others.
Group Session Rating Scale (GSRS) | Once per week for each session.
  The GSRS (Quirk et al., 2013) is a client-reported measure that assesses alliance, the quality of individual sessions, and helper skills.
Drexel University ACT/CT Adherence and Competence Rating Scale (DUACRS) | Once per week for each session.
  The DUACRS (McGrath, 2012) is a therapist-reported measure designed to assess adherence to CBT and ACT treatment components. While the original measure was designed to assess the extent to which each of these components occurred at every 5-minute interval during a session, we slightly adapted the response options to indicate whether the treatment components occurred at all in the relevant session.
California Psychotherapy Alliance Scale-Group- Therapist Version (CALPAS- G-TV) | Once per week for each session.
  The CALPAS-G-TV (Gaston & Marmar, 1994) is a therapist- report measure of the therapeutic alliance in group psychotherapy settings.
Clinical Global Impressions Scale (CGI) | Once per week for each session.
  The CGI (Guy, 1976) is a standard therapist-reported measure for making global assessments of clients' illness and improvement.
Chain of Change Ecological Momentary Assessment (ChaCha-EMA) | Three times per day for the seven days pre- and seven days post-treatment.
  The ChaCha-EMA consists of the same items assessed in the ChaCha-TD with the exception that questions will be phrased to assess clients' experiences at the moment of survey completion.

CONTACTS AND LOCATIONS:
Overall Officials: Iony D Ezawa, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dao A, Bernstein RA, Ramos FN, Beasley B, Ezawa ID. Unpacking the chain of change in group CBT and ACT for depression: A protocol for a randomized clinical trial. Contemp Clin Trials. 2025 Jun;153:107907. doi: 10.1016/j.cct.2025.107907. Epub 2025 Apr 2. PMID 40185199